CLINICAL TRIAL: NCT02902016
Title: Modulation of Lactase Expression by a New Synthetic PPARgamma Ligand in Ex-vivo Cultures of Duodenal Biopsies
Brief Title: Modulation of Lactase Expression by a New PPARgamma Ligand in Duodenal Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: French National Society of Gastroenterology (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013_68; 2015-A00259-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Lactose Intolerance
Keywords: PPARgamma; Lactose intolerance; Lactase
MeSH Terms: conditions — Lactose Intolerance; Carotid Intimal Medial Thickness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactase expression induction by GED (Experimental)
  Interventions: Drug: GED

INTERVENTIONS:
Drug: GED — Four duodenal biopsies will be collected. Two biopsies will stimulated with GED (PPARgamma modulator) ex vivo during 6 hours. Two biopsies will be unstimulated (control).

SUMMARY:
This study is designed to assess the effect of a new PPARgamma modulator on the expression and activity of the lactase enzyme in human intestinal epithelial cells. Based on their previous experimental results, the investigators hypothesized that modulating intestinal PPARgamma activity is a new pharmacological mechanism allowing the control of lactase expression and activity in the gut

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing gastroduodenal endoscopy for digestive cancer screening
* Subjects undergoing gastroduodenal endoscopy for ulcerative gastroduodenal diseases
* Subjects undergoing gastroduodenal endoscopy for epigastric pains
* Subjects undergoing gastroduodenal endoscopy for gastroesophageal reflux diseases

Exclusion Criteria:

* Subjects with macroscopic duodenal lesions detected at endoscopy
* Subjects suffering from coeliac disease
* Subjects suffering from atrophic gastritis
* Subjects who use anticoagulant
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
LCT mRNA expression measured by quantitative RT-PCR in duodenal biopsies stimulated ex-vivo with a new PPARgamma agonist (GED, 1mM) | 2 years

SECONDARY OUTCOMES:
LCT mRNA expression measured by quantitative RT-PCR in primary intestinal epithelial cells (isolated from duodenal biopsies) stimulated with a new PPARgamma agonist (GED, 1mM) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Desreumaux, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided